CLINICAL TRIAL: NCT03283254
Title: Preventing Postpartum Depression: A Dyadic Approach Adjunctive to Obstetric Care
Brief Title: PREPP: Preventing Postpartum Depression
Acronym: PREPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Catherine Monk, Diana Vagelos Professor of Women's Mental Health (in Obstetrics and Gynecology and Psychiatry), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAV4354; R01HD092062 (NIH); 7428 (Other: New York State Psychiatric Institute Institutional Review Board)
Record Dates: First submitted 2017-08-14; First posted 2017-09-14 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Depression (PPD)
Keywords: Postpartum Depression Treatment
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Two groups: One receives PREPP prevention intervention and the other group receives Enhanced Treatment as Usual (psychoeducation about Postpartum Depression, referral and monitoring)
Who Masked: Outcomes Assessor
Masking Description: The person administering the outcome measures is blind to participant group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practical Resources for Effective Postpartum (PREPP) (Experimental): A psychotherapeutic preventive intervention that involves psychoeducation and cognitive behavioral techniques.
  Interventions: Behavioral: Practical Resources for Effective Postpartum Parenting (PREPP)
- Enhanced Treatment as Usual (Active Comparator): Psychoeducation about Postpartum Depression, referral to treatment in the community and monitoring
  Interventions: Behavioral: Enhanced Treatment As Usual (ETAU)

INTERVENTIONS:
Behavioral: Practical Resources for Effective Postpartum Parenting (PREPP) — A preventive psychotherapy intervention for PPD: Participants in this arm of the study receive PREPP (Practical Resources for Effective Postpartum Parenting). PREPP is a brief preventive intervention for Postpartum Depression that focuses on the birthing parent-infant dyad and consists of 5 sessions that take place during pregnancy through 6 weeks postpartum carried out by study clinicians referred to as 'coaches.' The sessions of this preventive psychotherapy are comprised of three components: (a) mindfulness and self-reflection skills, (b) parenting skills and (c) psycho-education.
  Other Names: PREPP
  Arms: Practical Resources for Effective Postpartum (PREPP)
Behavioral: Enhanced Treatment As Usual (ETAU) — Psychoeducation, Clinical Assessment, Potential Referral: Participants receive "usual care" along with Postpartum Depression psychoeducation and enhanced support for finding perinatal mental healthcare treatment when appropriate by meeting with a study clinician specifically assigned to provide ETAU in this study at three times that are aligned with PREPP sessions that span from pregnancy to 6 weeks postpartum. At the first contact, participants meet with their assigned ETAU clinician and are given information about PPD, a brief clinical mental health assessment, and a referral for treatment if warranted or requested; the second session is a follow-up mental health clinical assessment with the study clinician and a referral for treatment if warranted or requested; at the third session, participants meet again with their study clinician and receive a mental health assessment, review relevant psychoeducation on PPD and are referred to treatment when appropriate.
  Other Names: ETAU
  Arms: Enhanced Treatment as Usual

SUMMARY:
The primary aim of this study is to determine if a behavioral intervention targeting maternal caregiving of young infants can increase infant sleep and reduce fuss/cry behavior, and thereby (1) reduce the incidence and/or severity of postpartum maternal depression and (2) improve the quality of the mother-infant interaction and subsequent child development. Specifically, the study team will investigate: (1) the effectiveness of the intervention compared to usual care; (2) if the effects of the intervention can be detected in the assessments of the quality of mother-infant interaction; (3) if there are prenatal and/or postnatal biomarkers that can help identify infants whose behavior is more likely to play a role in their mothers' depression; (4) if these markers differentiate which infants will be most responsive to the intervention(s); and (5), if assessments of brain function at birth and at 4-6 weeks of age provide biological nodal points for identifying the effects of the intervention on infant brain development. Participants will be recruited during their 2nd trimester, and will be randomly separated into one of two groups: a group that receives coaching in parenting techniques 3 coaching sessions and 2 check-in sessions or one that receives treatment as usual.

DETAILED DESCRIPTION:
Of the nearly 4 million mothers delivering live births each year in the United States, approximately 560,000 - or 14% - will develop major or minor depression within the first four months postpartum, when the rate peaks. This number dwarfs prevalence rates for gestational diabetes (2-5%) and is comparable to preterm birth (11.4%). Postpartum depression (PPD) has substantial consequences: poorer maternal quality of life, significant emotional suffering, and suicide risk. PPD predicts diminished mother-infant bonding, and poor outcomes in social-emotional and, in some groups, cognitive development. PPD is undertreated in part because women are reluctant to seek treatment due to the stigma associated with mental health care, logistical barriers to at-tending added health care appointments, and disinclination to take medications while breastfeeding. Of preventive interventions, few embed services in obstetrical care or leverage the unique mother-infant dyadic orientation of the childbearing period. The investigators developed a novel intervention based on the conceptualization of maternal depression as a potential disorder of the mother-infant dyad, and one that can be approached through psychological and behavioral changes in the mother - commencing before birth - that affect her and the child. PREPP (Practical Resources for Effective Postpartum Parenting) enrolls distressed pregnant women at risk for PPD, spans late pregnancy to the 6 week postpartum check up, comprises four in-person 'coaching' sessions adjunctive to obstetrical (OB) prenatal and postnatal appointments, one phone session, and imparts (a) mindfulness and self-reflection skills, (b) parenting skills, and (c) psycho-education.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women between 18-45 years old (based on self report)
2. A score of ≥19 on the Predictive Index of Postnatal Depression (PIPD), indicating risk for developing postpartum depression or score of ≥7 on the Edinburgh Postnatal Depression Scale
3. A healthy, singleton pregnancy (based on self report)
4. English speaking (based on self report)
5. Receiving standard prenatal care (based on self report)

Exclusion Criteria:

1. Multi-fetal pregnancy (based on self-report)
2. Smoking, illicit drug use, or alcohol use during pregnancy (based on self-report)
3. Acute medical illness or significant pregnancy complication (based on self-report)
4. Currently in weekly, individual psychotherapy, including psychopharmacology (based on self report)
5. Psychotic d/o; Bipolar I; Major Depressive d/o (based on M.I.N.I.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Monk, PhD, Principal Investigator — Columbia University; Elizabeth Werner, PhD, Study Director — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be made available to other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: After the completion of the study
Access Criteria: Permission of the PI

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only mothers were enrolled, and infants were assessed for efficacy
Groups:
- Practical Resources for Effective Postpartum (PREPP): Participants received the experimental PREPP intervention.
- Enhanced Treatment as Usual: Participants received enhanced treatment as usual (ETAU): Postpartum Depression psychoeducation, mood assessments, and referral for treatment if needed or requested by the participant.
Period: Overall Study
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Started | 88 | 87
6-week Postpartum Session | 69 | 66
12-week Postpartum Session | 52 | 52
16-week Postpartum Session | 57 | 57
Completed | 57 | 57
Not Completed | 31 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual | Total
Number analyzed (Participants) | 88 | 87 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.15 (5.51) | 30.16 (6.8) | 30.66 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 87 | 175
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 54 | 108
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 15 | 11 | 26
  White | 22 | 15 | 37
  More than one race | 7 | 3 | 10
  Unknown or Not Reported | 40 | 52 | 92
Region of Enrollment [Number; unit: participants]
  United States | 88 | 87 | 175

OUTCOME MEASURES:

1. Primary Outcome: Score on the Edinburgh Postnatal Depression Scale (EPDS)
Description: Maternal mood: Postpartum Depression Symptoms will be measured by Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a 10-item questionnaire that was developed to identify women who have postpartum depression. Items of the scale correspond to various clinical depression symptoms, such as guilt feeling, sleep disturbance, low energy, anhedonia, and suicidal ideation. Overall assessment is done by total score, which is determined by adding together the scores for each of the 10 items. Scores range from 0 to 30, with higher scores indicate more depressive symptoms (worse outcome).
Time Frame: Baseline, 6 weeks, 12 weeks, and 16 weeks postpartum
Population: Data for this outcome was only collected from participants who were able to attend a session to receive the intervention. Data was not collected from participants who did not attend a session.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 88 | 87
score on a scale
  Baseline | 5.04 (0.49) | 4.36 (3.51)
  6 week: number analyzed (Participants) | 69 | 66
  6 week | 4.43 (0.46) | 4.04 (0.42)
  12 week: number analyzed (Participants) | 52 | 52
  12 week | 3.51 (0.39) | 3.74 (0.42)
  16 week: number analyzed (Participants) | 57 | 57
  16 week | 3.69 (0.41) | 4.04 (0.44)

2. Primary Outcome: Score on the Pittsburgh Sleep Quality Index (PSQI)
Description: Maternal perception of sleep quality: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time interval. A total of 19 individual items generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Scores range from 0 to 21, where lower scores indicate a healthier sleep quality (better outcome).
Time Frame: Baseline, 6 weeks, 12 weeks, and 16 weeks postpartum
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 88 | 87
score on a scale
  Baseline | 7.01 (0.37) | 6.55 (0.35)
  6 week: number analyzed (Participants) | 69 | 66
  6 week | 7.21 (0.43) | 8.16 (0.47)
  12 week: number analyzed (Participants) | 52 | 52
  12 week | 5.73 (0.40) | 6.48 (0.44)
  16 week: number analyzed (Participants) | 57 | 57
  16 week | 5.88 (0.39) | 6.06 (0.40)

3. Primary Outcome: Score on HRSD-24
Description: The Hamilton Rating Scale for Depression (HRSD), also called the Hamilton Depression Rating Scale (HDRS), sometimes also abbreviated as HAM-D, is a multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. The patient is rated on 24 items scored either on a 3-point (0-2) or 5-point (0-4) Likert-type scale. Total scores range from 0 to 74 with a lower score indicating a better outcome.
Time Frame: Baseline, 6 weeks, 12 weeks, and 16 weeks postpartum
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 88 | 87
score on a scale
  Baseline | 4.09 (0.39) | 3.16 (0.32)
  6 week: number analyzed (Participants) | 69 | 66
  6 week | 3.23 (0.34) | 2.99 (0.32)
  12 week: number analyzed (Participants) | 52 | 52
  12 week | 2.99 (0.34) | 3.31 (0.37)
  16 week: number analyzed (Participants) | 57 | 57
  16 week | 2.74 (0.31) | 2.73 (0.31)

4. Primary Outcome: Score on the PHQ-9
Description: The nine-item Patient Health Questionnaire (PHQ-9) is a depressive symptom scale and diagnostic tool introduced in 2001 to screen adult patients in primary care settings. The instrument assesses for the presence and severity of depressive symptoms and a possible depressive disorder. It is scored by simply adding up the individual items' scores. Scores range from 0 to 27 with a lower score indicating a better outcome.
Time Frame: Baseline, 6 weeks, 12 weeks, and 16 weeks postpartum
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 88 | 87
score on a scale
  Baseline | 6.36 (0.49) | 5.64 (0.45)
  6 week: number analyzed (Participants) | 69 | 66
  6 week | 5.21 (0.44) | 5.42 (0.46)
  12 week: number analyzed (Participants) | 52 | 52
  12 week | 4.13 (0.39) | 5.19 (0.47)
  16 week: number analyzed (Participants) | 57 | 57
  16 week | 4.50 (0.41) | 4.08 (0.38)

5. Primary Outcome: Hamilton Anxiety Scale (HRSA)
Description: The scale consists of 14 items designed to assess the severity of a patient's anxiety. The patient is rated by on 14 items scored on a 5-point (0-4) Likert-type scale. Total scores range from 0 to 56 with a lower score indicating a better outcome.
Time Frame: Baseline, 6 weeks, 12 weeks, and 16 weeks postpartum
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 88 | 87
score on a scale
  Baseline | 4.09 (0.41) | 3.63 (0.37)
  6 week: number analyzed (Participants) | 69 | 66
  6 week | 3.01 (0.33) | 3.09 (0.34)
  12 week: number analyzed (Participants) | 52 | 52
  12 week | 3.01 (0.35) | 3.30 (0.38)
  16 week: number analyzed (Participants) | 57 | 57
  16 week | 2.93 (0.34) | 2.94 (0.34)

6. Primary Outcome: Sleep Efficiency (SEact) of the Mothers
Description: Sleep Efficiency (SEact) was measured by an activity monitor worn by the participants continuously over 7 days. SEact is reported as a percent of time spent asleep during the total time spent in bed.
Time Frame: 28-32 weeks gestation (prenatal), 34-39 weeks gestation (prenatal), 6 weeks postpartum, 16 weeks postpartum
Population: Data for this outcome could not be collected from participants who did not wear the activity monitor continuously for 7 days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 25 | 29
percent
  28-32 weeks gestation | 71.90 (21.25) | 73.44 (25.21)
  34-39 weeks gestation: number analyzed (Participants) | 19 | 22
  34-39 weeks gestation | 74.00 (22.67) | 71.28 (24.31)
  6 week postpartum: number analyzed (Participants) | 12 | 12
  6 week postpartum | 65.32 (25.55) | 71.14 (20.78)
  16 week postpartum: number analyzed (Participants) | 8 | 7
  16 week postpartum | 69.25 (22.24) | 76.74 (17.91)

7. Secondary Outcome: Total Nocturnal Sleep Duration - Brief Infant Sleep Questionnaire (BISQ)
Description: The BISQ is a parent-reported questionnaire on infants/toddler (0-29 months) sleep over 7 days
Time Frame: 6 weeks and 16 weeks postpartum
Population: Data was not collected from participants who did not complete this measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 63 | 64
hours
  6 weeks | 7.27 (2.08) | 7.26 (1.97)
  16 weeks: number analyzed (Participants) | 50 | 55
  16 weeks | 8.24 (2.12) | 8.30 (1.79)

8. Secondary Outcome: Total Daytime Sleep Duration - Brief Infant Sleep Questionnaire (BISQ)
Description: The BISQ is a parent-reported questionnaire on infants/toddler (0-29 months) sleep over 7 days.
Time Frame: 6 weeks and 16 weeks postpartum
Population: Data was not collected from participants who did not complete this measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 63 | 64
hours
  6 weeks | 6.17 (2.66) | 6.65 (2.47)
  16 weeks: number analyzed (Participants) | 52 | 57
  16 weeks | 4.84 (2.45) | 4.50 (1.87)

9. Secondary Outcome: Total Number of Instances of Waking up at Night - Brief Infant Sleep Questionnaire (BISQ)
Description: The BISQ is a parent-reported questionnaire on infants/toddler (0-29 months) sleep over 7 days.
Time Frame: 6 weeks and 16 weeks postpartum
Population: Data was not collected from participants who did not complete this measure.
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 63 | 64
awakenings
  6 weeks | 2.61 (1.05) | 2.71 (1.17)
  16 weeks: number analyzed (Participants) | 52 | 57
  16 weeks | 1.77 (1.08) | 1.85 (1.26)

10. Secondary Outcome: Total Settling Time to Fall Asleep for the Night - Brief Infant Sleep Questionnaire (BISQ)
Description: The BISQ is a parent-reported questionnaire on infants/toddler (0-29 months) sleep over 7 days.
Time Frame: 6 weeks and 16 weeks postpartum
Population: Data was not collected from participants who did not complete this measure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 62 | 62
minutes
  6 weeks | 41.23 (35.04) | 31.35 (20.16)
  16 weeks: number analyzed (Participants) | 52 | 56
  16 weeks | 31.21 (22.50) | 32.23 (30.07)

11. Secondary Outcome: Daily Minutes of Infant Crying Over 4 Days
Description: Cry behavior will be measured by The Baby Day Diary, which is a 24-hour diary of infant and parental behavior for days. The number of minutes for the crying behavior is averaged over a span of 4 days, with a higher number indicating a worse outcome.
Time Frame: 6 weeks and 16 weeks postpartum
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 88 | 87
minutes per day
  6 weeks | 164.72 (81.32) | 117.35 (72.46)
  16 weeks | 98.75 (66.58) | 101.25 (48.23)

12. Secondary Outcome: Length of Longest Sleep at Night for Infants Over 4 Days
Description: Sleep behavior will be measured by The Baby Day Diary, which is a 24-hour diary of infant and parental behavior for days. The number of minutes of sleep is averaged over a span of 4 days. A higher number indicates a better outcome.
Time Frame: 6 weeks and 16 weeks postpartum
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 88 | 87
minutes
  6 weeks | 249.52 (81.04) | 238.24 (106.78)
  16 weeks | 291.52 (71.91) | 277.67 (74.33)

13. Secondary Outcome: Total Sleep Time (TSTact) in the Mothers
Description: TSTact was measured by an activity monitor worn by the participants continuously over 7 days.
Time Frame: 28-32 weeks gestation (prenatal), 34-39 weeks gestation (prenatal), 6 weeks postpartum, 16 weeks postpartum
Population: Data for this outcome was not collected from participants who did not wear the activity monitor continuously for 7 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 25 | 29
minutes
  28-32 weeks gestation | 305.03 (163.77) | 291.34 (180.48)
  34-39 weeks gestation: number analyzed (Participants) | 19 | 22
  34-39 weeks gestation | 329.17 (168.50) | 274.50 (170.60)
  6 weeks postpartum: number analyzed (Participants) | 12 | 12
  6 weeks postpartum | 273.89 (159.13) | 249.66 (161.42)
  16 weeks postpartum: number analyzed (Participants) | 8 | 7
  16 weeks postpartum | 282.90 (152.18) | 286.00 (141.96)

14. Other Pre Specified Outcome: Total Daily Minutes of Sleep Reported on the Self-Reported Sleep Log (Mother)
Description: Self-reported sleep time was recorded by participants each night over a span of 7 days.
Time Frame: 28-32 weeks gestation (prenatal), 34-39 weeks gestation (prenatal), 6 weeks postpartum, 16 weeks postpartum
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
Number analyzed (Participants) | 88 | 87
minutes per day
  28-32 weeks gestation | 393.51 (72.90) | 402.90 (78.21)
  34-39 weeks gestation | 394.25 (97.37) | 390.10 (92.38)
  6 weeks postpartum | 370.01 (125.64) | 336.02 (75.83)
  16 weeks postpartum | 408.90 (91.20) | 381.45 (72.54)

ADVERSE EVENTS:
Time Frame: During each assessment session, from 20-29 weeks gestation to 16 weeks postpartum, approximately 21- 36 weeks of participation
Arm/Group | Practical Resources for Effective Postpartum (PREPP) | Enhanced Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/87
Other Adverse Events (participants affected / at risk) | 0/88 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT03283254/Prot_SAP_000.pdf